CLINICAL TRIAL: NCT00878306
Title: Disulfiram Interactions With HIV Medications: Clinical Implications
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None
Other Study IDs: R01DA024982 (NIH); R01DA024982 (NIH)
Record Dates: First submitted 2009-04-07; First posted 2009-04-08 (Estimated); Last update posted 2014-05-06 (Estimated); Status verified 2014-05

CONDITIONS: HIV Infections; Drug Abuse
Keywords: Treatment of drug dependency with HIV medications; HIV
MeSH Terms: conditions — HIV Infections; Substance-Related Disorders | interventions — Disulfiram; efavirenz; Atazanavir Sulfate; Ritonavir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Disulfiram (Active Comparator): Disulfiram
  Interventions: Drug: Disulfiram
- Disulfiram + Efavirenz (Experimental): Efavirenz alone, then in addition with Disulfiram
  Interventions: Drug: Disulfiram + Efavirenz
- Disulfiram + Atazanavir (Experimental): Atazanavir alone, then in addition with Disulfiram
  Interventions: Drug: Disulfiram + Atazanavir
- Disulfiram + Ritonavir (Experimental): Ritonavir alone, then in addition with Disulfiram
  Interventions: Drug: Disulfiram + Ritonavir

INTERVENTIONS:
Drug: Disulfiram — 62.5 mg daily x3 days, then 250 mg daily x3 days
  Other Names: Antabuse
  Arms: Disulfiram
Drug: Disulfiram + Efavirenz — Efavirenz 600 mg daily x10 days, then in addition with 62.5 mg daily x3 days, then Disulfiram 250 mg daily x3 days
  Arms: Disulfiram + Efavirenz
Drug: Disulfiram + Atazanavir — Atazanavir 400 mg daily x8 days, then in addition with 62.5 mg daily x3 days, then Disulfiram 250 mg daily x3 days
  Arms: Disulfiram + Atazanavir
Drug: Disulfiram + Ritonavir — Ritonavir 200 mg daily x8 days, then in addition with 62.5 mg daily x3 days, then Disulfiram 250 mg daily x3 days
  Arms: Disulfiram + Ritonavir

SUMMARY:
The purpose of this study is to determine whether disulfiram might be a safe and effective treatment for cocaine and/or alcohol dependence in patients with HIV disease. This research is designed to characterize the presence or absence of significant drug interactions between disulfiram and HIV medications using standard clinical pharmacology techniques as well as monitor any side effects that might occur when these medications are administered together.

DETAILED DESCRIPTION:
Cocaine and alcohol abuse are strongly linked to HIV infection and transmission of the virus. Disulfiram has long been approved by the US FDA for the treatment of alcohol and recent data shows it to be effective in reducing cocaine abuse. Disulfiram and antiretroviral medications (ARV) are metabolized by cytochrome P450 3A and concomitant use of these drugs could potentially produce adverse drug interactions underscoring the need to identify and understand the clinical implications of these drug interactions in order to more effectively treat individuals with both HIV disease and cocaine and/or alcohol use disorders. This will be accomplished by conducting studies aimed at identifying whether pharmacokinetic or pharmacodynamic drug interactions of importance occur between disulfiram and medications frequently utilized in those with HIV/AIDS.

Abuse of cocaine and/or alcohol has been shown to be a significant risk factor for HIV infections as a result of high risk sexual and drug use behaviors occurring in the context of use of these substances. Those with HIV infection and untreated cocaine and/or alcohol dependence are also at a high risk of transmitting HIV to others. Moreover, those with HIV disease and substance dependence often experience poor clinical outcomes as a result of nonadherence to HIV treatment regimens.

Disulfiram (DIS) is an inhibitor of ALDH and has been reported to alter hepatic cytochrome P450 enzyme function important to metabolism of many drugs frequently used in the treatment of HIV/AIDS. Although approved for the treatment of alcohol dependence, DIS has been studied as a treatment for cocaine addiction in recent years. DIS at the standard 250 mg daily dose has been associated with significant reductions in cocaine use as well as alcohol use in those with histories of concomitant cocaine-alcohol abuse. DIS 250 mg daily has been shown to have a significant pharmacokinetic interaction with cocaine resulting in delayed cocaine clearance. In order to more fully access possible use of DIS treatment for cocaine and/or alcohol dependence in this population, it is important to determine if any excess risk is conveyed as a result of drug interactions that might occur between DIS and the ARV medications.

This study will be using a standard clinical pharmacology study design using a within-subject design examining the two drug interaction studies between DIS (250 mg daily) and the following medications:

1. Non-nucleoside reverse transcriptase inhibitor, efavirenz 600 mg daily for 10 days
2. Protease inhibitors atazanavir 400 mg daily for 8 days or ritonavir 200 mg daily for 8 days

   Additional data will be collected and analyzed including:
3. Clinical data on effects of these medications alone and in combination on cardiac conduction, hepatic function, and serum lipids will be obtained
4. The safety of co-administration of alcohol containing HIV preparations (ritonavir) with DIS will be determined
5. The effect of ARV on DIS function as determined by ALDH activity and DIS and metabolite concentrations will be determined using a control sample within-subject design (DIS doses of 62.5 mg and 250 mg daily) and between subjects design.

ELIGIBILITY:
Inclusion Criteria:

* Good health and without clinical findings that require medical or psychiatric intervention as determined by a physical and mental status examination and screening laboratory tests, urinalysis, and ECG
* 18 years of age or older
* Willing to abstain from alcohol during the study and for two weeks afterward

Exclusion Criteria:

* Patients who are receiving concurrently other drugs that are inducers or inhibitors of hepatic microsomal enzymes
* Patients with a known sensitivity to the HIV therapeutics to be studied
* Pregnant or nursing mothers
* Current major affective or psychotic illnesses or suicidality
* Clinically active hepatitis
* Diabetes, hyperlipidemia, coagulation disorders, or renal disease will be excluded
* Those meeting criteria for current alcohol or drug dependence (other than nicotine)
* HIV infection

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2008-11; Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
The effect of disulfiram on the pharmacokinetics of each of the antiretroviral medications to be studied | Measured at Day 15

SECONDARY OUTCOMES:
The effect of the antiretroviral medications on disulfiram measured by ALDH activity and disulfiram pharmacokinetics | Measured at Day 0, Day 4, and Day 8
Cardiac Conduction | Measured at screening and during pharmacokinetic studies
Hepatic Function | Measured at screening and during pharmacokinetic studies
Serum Lipids | Measured at screening and during pharmacokinetic studies
Safety of co-administration of alcohol containing HIV preparations (ritonavir) and Disulfiram | Measured at day 11- day 15

CONTACTS AND LOCATIONS:
Overall Officials: Elinore F McCance-Katz, M.D., Ph.D, Principal Investigator — University of California, San Francisco
Locations (1):
- San Francisco General Hospital, San Francisco, California, United States